CLINICAL TRIAL: NCT07382037
Title: Efficacy of Whole-Body Vibration in Patients With Patellofemoral Pain Syndrome: A Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Whole-Body Vibration in Patients With Patellofemoral Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Hakan Alkan, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PamukkaleU.ftr-HAlkan-001
Record Dates: First submitted 2025-08-09; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: Patellofemoral Pain, PFP
Keywords: whole body vibration; knee
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Whole body vibration group, 3 days a week, 30 minutes a day for 8 weeks
  Interventions: Device: Whole body vibration
- Sham group (Sham Comparator): Sham-whole body vibration, 3 days a week, 30 minutes a day for 8 weeks
  Interventions: Device: Sham Whole Body Vibration

INTERVENTIONS:
Device: Whole body vibration — In this group, prior to the patient stepping onto the platform, the practitioner will turn off the vibration motor of the device and activate an external motor (which is not in contact with the WBV device, has no effective vibration capability, and only produces sound), installed by our team. Since the visual display of the device remains active, patients will not be aware that the actual vibration function is disabled, thereby preventing any bias related to device inactivity.
  Arms: Experimental
Device: Sham Whole Body Vibration — In this group, prior to the patient stepping onto the platform, the practitioner will turn off the vibration motor of the device and activate an external motor (which is not in contact with the WBV device, has no effective vibration capability, and only produces sound), installed by our team. Since the visual display of the device remains active, patients will not be aware that the actual vibration function is disabled, thereby preventing any bias related to device inactivity.
  Arms: Sham group

SUMMARY:
Patellofemoral Pain Syndrome (PFPS), or anterior knee pain, is one of the most common disorders affecting the lower extremities.

Currently, there is no established "gold standard" treatment for PFPS. However, various interventions-including strengthening of the hip and knee muscles (e.g., hip abductors, external rotators, and knee extensors), taping, bracing, foot orthoses, manual therapy, acupuncture, blood flow restriction training, and conventional physical agents (e.g., ultrasound, cryotherapy, neuromuscular electrical stimulation, laser therapy, electromyographic biofeedback, etc.)-have been reported to provide meaningful clinical benefits. Strengthening of the hip and knee muscles alone has been shown to improve both pain and function in the short, medium, and long term. In recent high-quality studies, hip and knee muscle strengthening has been recognized as an effective "classical" treatment approach for PFPS. Regarding the mechanism of pain relief, previous research suggests that strengthening these muscles may alleviate pain by stabilizing patellar motion and/or reducing pressure on the patellofemoral joint.

Similar to traditional resistance training, whole-body vibration (WBV) training is an alternative method for muscle strengthening. WBV platforms can generate vertical vibrations that stimulate tonic vibration reflexes through muscle spindles, thereby activating homonymous alpha motor neurons and inducing reflex muscle contractions. As a result, increased motor unit recruitment enhances the excitability of muscle spindles, leading to improved muscle strength. Additionally, WBV training can improve muscle balance, strength, and function. Therefore, combining WBV with hip and knee strengthening exercises may represent a more effective treatment strategy for PFPS. The aim of this study is to evaluate whether the combination of WBV and hip-knee muscle strengthening is more effective in reducing pain and improving function than hip-knee strengthening alone.

DETAILED DESCRIPTION:
Patellofemoral Pain Syndrome (PFPS), or anterior knee pain, is one of the most common disorders affecting the lower extremities.

Currently, there is no established "gold standard" treatment for PFPS. However, various interventions-including strengthening of the hip and knee muscles (e.g., hip abductors, external rotators, and knee extensors), taping, bracing, foot orthoses, manual therapy, acupuncture, blood flow restriction training, and conventional physical agents (e.g., ultrasound, cryotherapy, neuromuscular electrical stimulation, laser therapy, electromyographic biofeedback, etc.)-have been reported to provide meaningful clinical benefits. Strengthening of the hip and knee muscles alone has been shown to improve both pain and function in the short, medium, and long term. In recent high-quality studies, hip and knee muscle strengthening has been recognized as an effective "classical" treatment approach for PFPS. Regarding the mechanism of pain relief, previous research suggests that strengthening these muscles may alleviate pain by stabilizing patellar motion and/or reducing pressure on the patellofemoral joint.

Similar to traditional resistance training, whole-body vibration (WBV) training is an alternative method for muscle strengthening. WBV platforms can generate vertical vibrations that stimulate tonic vibration reflexes through muscle spindles, thereby activating homonymous alpha motor neurons and inducing reflex muscle contractions. As a result, increased motor unit recruitment enhances the excitability of muscle spindles, leading to improved muscle strength. Additionally, WBV training can improve muscle balance, strength, and function. Therefore, combining WBV with hip and knee strengthening exercises may represent a more effective treatment strategy for PFPS. The aim of this study is to evaluate whether the combination of WBV and hip-knee muscle strengthening is more effective in reducing pain and improving function than hip-knee strengthening alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years,
* Diagnosed with unilateral Patellofemoral Pain Syndrome (PFPS),
* Reporting anterior knee pain or pain behind the patella in at least two of the following activities:

ascending stairs, jumping, running, squatting, kneeling, prolonged sitting,

- Positive results in at least two of the following clinical tests: Eccentric step-down test, Patellar border tenderness test, Patellar grind (Clarke's) or apprehension test,

* Ability to understand the procedures, potential benefits, and possible adverse effects,
* Willingness to participate in the treatment program.

Exclusion Criteria:

* Severe injury or pathological changes in knee structures (e.g., ligaments, menisci, patellar tendons, iliotibial bands, joint capsules, or plicae),
* History of significant trauma or surgery involving the knee or lower extremity,
* History of patellar dislocation or subluxation,
* Diagnosis of Osgood-Schlatter disease or Sinding-Larsen-Johansson syndrome,
* Joint effusion in the knee, or presence of redness, swelling, or increased warmth on physical examination,
* Serious systemic conditions, including cardiovascular diseases, tumors, gallstones or kidney stones, severe disc or spinal lesions, pacemaker implantation, epilepsy, recent fractures or surgeries, or acute arthritis,
* Pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
VAS | Change from baseline VAS at the 8th week after the treatment
  Pain is the most characteristic symptom in Patellofemoral Pain Syndrome (PFPS). After recording the duration of pain (in months) for each patient, pain intensity was assessed using the Visual Analog Scale (VAS), which is a 10-centimeter (cm) line anchored by 0 (no pain) and 10 (unbearable pain). Patients were asked to rate their pain at rest, during stair ascent/descent, squatting, prolonged sitting, and walking. Crossley et al. have reported that the VAS is a valid, reliable, and responsive tool for assessing pain in individuals with PFPS

SECONDARY OUTCOMES:
Anterior Knee Pain Scale | Change from baseline AKPS score at the 8th week after the treatment
  Subjective symptoms and functional limitations of patients with Patellofemoral Pain Syndrome (PFPS) were evaluated using the Kujala Patellofemoral Scoring System. This scoring system was developed by Kujala et al. in 1993, and it allows for functional assessment of knee pathologies related to the patellofemoral structure. The Kujala Patellofemoral Pain Score consists of 13 subcategories evaluating limping, weight bearing, walking, stair activities, squatting, jumping, prolonged sitting with knees flexed at 90°, running, pain, swelling, abnormal painful patellar movement, thigh atrophy, and loss of flexion. The total score ranges from 0 to 100 points, with 100 indicating the best functional status.
Short Form - 36 | Change from baseline SF-36 score at the 8th week after the treatment
  The quality of life of all patients will be assessed using the Short Form-36 Health Survey (SF-36). This instrument consists of 36 items and measures eight health domains:
  Physical functioning (10 items), Social functioning (2 items), Role limitations due to physical problems (4 items), Role limitations due to emotional problems (3 items), Mental health (5 items), Energy/vitality (4 items), Bodily pain (2 items), and General health perception (5 items)
Muscle Mass Assessment via Ultrasound | Change from baseline muscle mass assessment at the 8th week after the treatment
  Muscle mass measurements of the vastus medialis and gluteus medius muscles will be performed using ultrasound (Clarius™ by Clarius Mobile Health) both before and after treatment.
  For the vastus medialis, the patient will be positioned supine with the knee in approximately 30 degrees of flexion. The ultrasound probe will be placed on the medial quadriceps region, between the medial border of the patella and the medial femoral condyle. The probe will be angled at approximately 45° to the long axis of the femur, oriented parallel to the muscle fibers.
  For the gluteus medius, the patient will be positioned in side-lying, with the painful side facing upward. The probe will be placed at the lower half of the distance between a line connecting the anterior superior iliac spine (ASIS) and the posterior superior iliac spine (PSIS) and the greater trochanter.
  Measurements will be performed by the same evaluator at baseline and at the 8th week following treatment.
Change in peak torque at 60°/s (Nm) of the knee muscles measured by isokinetic dynamometer | Change from baseline to Week 8 after treatment
  Isokinetic assessment of the symptomatic (painful) knee will be performed using the IsoMed 2000 Isokinetic System. Participants will be seated in an upright position with stabilization of the trunk and lower limbs. Peak Torque (PT, measured in Newton-meters, Nm) represents the maximum torque generated during knee flexion and extension at an angular velocity of 60°/s. Participants will perform four maximal repetitions following three familiarization trials. The change in PT from baseline to week 8 will be used to assess improvement in knee muscle endurance at higher movement speeds.
Change in peak torque at 240°/s (Nm) of the knee muscles measured by isokinetic dynamometer | Change from baseline to Week 8 after treatment
  Isokinetic assessment of the symptomatic (painful) knee will be performed using the IsoMed 2000 Isokinetic System. Participants will be seated in an upright position with stabilization of the trunk and lower limbs.
  Peak Torque (PT, measured in Newton-meters, Nm) represents the maximum torque generated during knee flexion and extension at an angular velocity of 240°/s. Participants will perform ten maximal repetitions following three familiarization trials.
  The change in PT from baseline to week 8 will be used to assess improvement in knee muscle endurance at higher movement speeds.
Assessment of the hamstring/quadriceps ratio at 60°/s with an isokinetic dynamometer | Change from baseline VAS at the 8th week after the treatment
  The H/Q ratio will be calculated using the peak torque values obtained from the isokinetic tests at 60°/s.
  Specifically, it is determined by dividing the hamstring peak torque by the quadriceps peak torque measured during the same test session.
  The H/Q ratio at this slower speed reflects the strength balance between the knee flexors and extensors under controlled movement conditions.
  A balanced ratio is crucial for joint stability and injury prevention, particularly in patients with knee pain or dysfunction.
  Testing will be conducted using the IsoMed 2000, with the patient's position and stabilization identical to other isokinetic assessments.
Assessment of the hamstring/quadriceps ratio at 240°/s with an isokinetic dynamometer | Change from baseline to week 8 after treatment
  The H/Q ratio will also be calculated at 240°/s, based on the peak torque values obtained from the high-velocity isokinetic test.
  It is computed by dividing the hamstring peak torque by the quadriceps peak torque at this higher angular velocity.
  The H/Q ratio at 240°/s assesses the dynamic balance and neuromuscular coordination between flexor and extensor muscle groups during rapid movements.
  Maintaining an appropriate H/Q ratio at faster speeds is considered an important indicator of functional knee stability and injury resilience.
  All procedures (positioning, stabilization, familiarization, and repetitions) will be performed identically to the other isokinetic test conditions, using the IsoMed 2000 system.
Change in Total Work (J) of the Knee Muscles at 60°/s With an Isokinetic Dynamometer | Change from baseline to Week 8 after treatment
  Isokinetic assessments of the symptomatic (painful) knee will be performed using the IsoMed 2000 Isokinetic System. Participants will be seated in an upright position, with the chest, waist, and lower limbs secured to ensure proper body stabilization and minimize compensatory movements.
  To obtain reliable data on muscle performance, testing at an angular velocity of 60°/s will include four consecutive maximal concentric repetitions of knee flexion and extension. Prior to the test, participants will perform three familiarization repetitions at the same velocity to become accustomed to the movement and the device.
  Total Work (TW), measured in Joules (J), represents the total amount of work performed by the knee flexor and extensor muscles across all repetitions at 60°/s.
  This parameter reflects overall muscular endurance and energy output of the quadriceps and hamstrings during slower, controlled movements.
Change in Total Work (J) of the Knee Muscles at 240°/s With an Isokinetic Dynamometer | Change from baseline to Week 8 after treatment
  Isokinetic assessments of the symptomatic (painful) knee will be conducted using the IsoMed 2000 Isokinetic System. Participants will be positioned in an upright seated position, and the chest, waist, and lower limbs will be secured with straps to ensure body stabilization during testing.
  For this evaluation, an angular velocity of 240°/s will be used, and patients will perform ten consecutive maximal concentric repetitions of knee flexion and extension. Before the test, three familiarization repetitions at the same angular velocity will be completed to ensure accurate and consistent performance.
  Total Work (TW), expressed in Joules (J), will represent the total energy output of the knee flexor and extensor muscles during all repetitions at 240°/s.
  This measurement provides information on muscular endurance, power, and performance efficiency of the knee muscles under high-velocity dynamic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Alkan, Prof Dr, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dag F, Dal U, Altinkaya Z, Erdogan AT, Ozdemir E, Yildirim DD, Colak M. Alterations in energy consumption and plantar pressure distribution during walking in young adults with patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2019 Jan;53(1):50-55. doi: 10.1016/j.aott.2018.10.006. Epub 2018 Oct 25. PMID 30482589
- [Background] Corum M, Basoglu C, Yakal S, Sahinkaya T, Aksoy C. Effects of whole body vibration training on isokinetic muscular performance, pain, function, and quality of life in female patients with patellofemoral pain: a randomized controlled trial. J Musculoskelet Neuronal Interact. 2018 Dec 1;18(4):473-484. PMID 30511951
- [Background] Dieterich AV, Pickard CM, Strauss GR, Deshon LE, Gibson W, McKay J. Muscle thickness measurements to estimate gluteus medius and minimus activity levels. Man Ther. 2014 Oct;19(5):453-60. doi: 10.1016/j.math.2014.04.014. Epub 2014 May 10. PMID 24880207
- [Background] Dogan A, Sengul I, Askin A, Tosun A. Effect of static knee joint flexion on vastus medialis obliquus fiber angle in patellofemoral pain syndrome: An ultrasonographic study. PM R. 2022 Jul;14(7):802-810. doi: 10.1002/pmrj.12655. Epub 2021 Jul 23. PMID 34165244
- [Background] Kuru T, Dereli EE, Yaliman A. Validity of the Turkish version of the Kujala patellofemoral score in patellofemoral pain syndrome. Acta Orthop Traumatol Turc. 2010;44(2):152-6. doi: 10.3944/AOTT.2010.2252. PMID 20676018
- [Background] Kujala UM, Jaakkola LH, Koskinen SK, Taimela S, Hurme M, Nelimarkka O. Scoring of patellofemoral disorders. Arthroscopy. 1993;9(2):159-63. doi: 10.1016/s0749-8063(05)80366-4. PMID 8461073
- [Background] Takanashi Y, Chinen Y, Hatakeyama S. Whole-body vibration training improves the balance ability and leg strength of athletic throwers. J Sports Med Phys Fitness. 2019 Jul;59(7):1110-1118. doi: 10.23736/S0022-4707.18.09012-6. Epub 2018 Oct 10. PMID 30317837
- [Background] Alam MM, Khan AA, Farooq M. Effect of whole-body vibration on neuromuscular performance: A literature review. Work. 2018;59(4):571-583. doi: 10.3233/WOR-182699. PMID 29733043
- [Background] Petersen W, Rembitzki I, Liebau C. Patellofemoral pain in athletes. Open Access J Sports Med. 2017 Jun 12;8:143-154. doi: 10.2147/OAJSM.S133406. eCollection 2017. PMID 28652829
- [Background] Crossley KM, Callaghan MJ, van Linschoten R. Patellofemoral pain. Br J Sports Med. 2016 Feb;50(4):247-50. doi: 10.1136/bjsports-2015-h3939rep. PMID 26834209
- [Background] Ho KY, Keyak JH, Powers CM. Comparison of patella bone strain between females with and without patellofemoral pain: a finite element analysis study. J Biomech. 2014 Jan 3;47(1):230-6. doi: 10.1016/j.jbiomech.2013.09.010. Epub 2013 Oct 15. PMID 24188973
- [Background] Cheung RT, Zhang Z, Ngai SP. Different relationships between the level of patellofemoral pain and quality of life in professional and amateur athletes. PM R. 2013 Jul;5(7):568-72. doi: 10.1016/j.pmrj.2012.12.007. Epub 2013 Jan 29. PMID 23375635
- [Background] Smith BE, Selfe J, Thacker D, et al. Incidence and prevalence of patellofemoral pain: a systematic review and meta-analysis. PLoS One. 2018;13(1):e0190892.
- [Background] Dey P, Callaghan M, Cook N, et al. A questionnaire to identify patellofemoral pain in the community: an exploration of measurement properties. BMC Musculoskelet Disord. 2016;17:237.
- [Background] Willy RW, Hoglund LT, Barton CJ, Bolgla LA, Scalzitti DA, Logerstedt DS, et al. Patellofemoral pain: clinical practice guidelines linked to the International Classification of Functioning, Disability and Health from the Academy of Orthopaedic Physical Therapy of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2019;49(9):CPG1-CPG95.